CLINICAL TRIAL: NCT02109133
Title: The Impacts of Surgical Visibility Through Deep Neuromuscular Blockade on Intraocular Pressure in Patients Undergoing Robot-Assisted Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2014-0058
Record Dates: First submitted 2014-03-30; First posted 2014-04-09 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Robot-Assisted Laparoscopic Radical Prostatectomy
Keywords: deep neuromuscular blockade; intraocular pressure
MeSH Terms: interventions — Rocuronium; Sugammadex; Atracurium; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep neuromuscular blockade (Experimental): Deep neuromuscular blockade
  Interventions: Procedure: deep neuromuscular blockade; Drug: Rocuronium; Drug: Sugammadex
- moderate neuromuscular blockade (Active Comparator): moderate neuromuscular blockade
  Interventions: Procedure: moderate neuromuscular blockade; Drug: Atracurium; Drug: Neostigmine

INTERVENTIONS:
Procedure: deep neuromuscular blockade — deep neuromuscular blockade using rocuronium and reverse with sugammadex
  Arms: Deep neuromuscular blockade
Procedure: moderate neuromuscular blockade — moderate neuromuscular blockade using atracurium and reverse with neostigmine
  Arms: moderate neuromuscular blockade
Drug: Rocuronium
  Arms: Deep neuromuscular blockade
Drug: Sugammadex
  Arms: Deep neuromuscular blockade
Drug: Atracurium
  Arms: moderate neuromuscular blockade
Drug: Neostigmine
  Arms: moderate neuromuscular blockade

SUMMARY:
Intraocular pressure is significantly increase during robot-assisted laparoscopic radical prostatectomy which is performed in a steep trendelenburg position at prolonged times of pneumoperitoneum. Therefore investigators decided to evaluate the impacts of surgical visibility through deep neuromuscular blockade on intraocular pressure in patients undergoing Robot-Assisted Laparoscopic Radical Prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-II
2. obtaining written informed consent from the parents
3. aged over 50 years who were undergoing robot- assisted laparoscopic prostatectomy

Exclusion Criteria:

1. eye surgery previously
2. unstable angina or congestive heart failure
3. concomitant eye disease (glaucoma, diabetic retinopathy, cataract, retinal detachment)
4. high intraocular pressure over 30mmHg after screening test.
5. uncontrolled hypertension (diastolic bp>110mmHg)
6. coagulopathy
7. asthma
8. hepatic failure
9. renal failure(creatinine clearance < 30 ml/min)
10. drug hyperactivity
11. neurological or psychiatric illnesses
12. mental retardation
13. patients who can't read the consent form due to illiterate or foreigner
14. previous malignant hyperthermia Hx
15. drug medication which interact with muscle relaxant (anti-convulsant, certain antibiotics, magnesium etc)
16. BMI > 30kg/m2

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Yoo YC, Kim NY, Shin S, Choi YD, Hong JH, Kim CY, Park H, Bai SJ. The Intraocular Pressure under Deep versus Moderate Neuromuscular Blockade during Low-Pressure Robot Assisted Laparoscopic Radical Prostatectomy in a Randomized Trial. PLoS One. 2015 Aug 28;10(8):e0135412. doi: 10.1371/journal.pone.0135412. eCollection 2015. PMID 26317357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 1 site in the Korea
Pre-assignment Details: No test entered
Groups:
- Moderate Neuromuscular Blockade (Moderate NMB Group): Moderate NMB Group included patients who received an IV atracurium bolus (0.5 mg kg-1) following the continuous infusion of 0.3 mg kg-1 until the end of the ST position. Dose titration was assigned to an attending anaesthetist via regulation of the bolus infusion speed to maintain a TOF count of 1 to 2. Neostigmine was used to reverse the effects of NMB after surgery.
- Deep Neuromuscular Blockade (Deep NMB Group): Deep NMB Group included patients who received an intravenous (IV) rocuronium bolus (1.0 mg kg-1) following the continuous infusion of 0.6 mg kg-1 until the end of the ST position. Dose titration was assigned to an attending anaesthetist via regulation of the bolus infusion speed to maintain a post-tetanic count (PTC) of 1 to 2. Sugammadex was administered to reverse the effects of NMB after surgery.
Period: Overall Study
Arm/Group | Moderate Neuromuscular Blockade (Moderate NMB Group) | Deep Neuromuscular Blockade (Deep NMB Group)
Started | 33 | 34
Completed | 32 | 34
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moderate Neuromuscular Blockade: moderate neuromuscular blockade: moderate neuromuscular blockade using atracurium and reverse with neostigmine
  Atracurium
  Neostigmine
- Deep Neuromuscular Blockade: deep neuromuscular blockade: deep neuromuscular blockade using rocuronium and reverse with sugammadex
  Rocuronium
  Sugammadex
- Total: Total of all reporting groups
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 22 | 38
  >=65 years | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.1) | 61.5 (5.4) | 62.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 34 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 32 | 34 | 66
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Maximum Intraocular Pressure During RALRP Under Deep Neuromuscular Blockade
Description: maximum intraocular pressure during RALRP under deep neuromuscular blockade after being positioned in the steep Trendelenburg position with CO2 pneumoperitoneum under deep neuromuscular blockade
Time Frame: Maximum intraocular pressure was measured at 60 minutes after CO2 pneumoperitoneum in the ST position
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Moderate Neuromuscular Blockade (Moderate NMB Group) | Deep Neuromuscular Blockade (Deep NMB Group)
Number analyzed (Participants) | 32 | 34
mmHg | 23.3 (2.7) | 19.8 (2.1)

2. Secondary Outcome: Overall Surgical Condition
Description: overall surgical conditions using the 5-point rating scale as previously described: Grade 5 (optimal), optimal surgical conditions; grade 4 (good), nonoptimal conditions, but an intervention is not required; grade 3 (acceptable), wide surgical view, but an intervention can improve surgical conditions, grade 2 (poor), inadequate conditions, there is a visible view, but an intervention is necessary to ensure acceptable surgical conditions; grade 1 (extremely poor), inability to perform surgery; therefore, intervention is necessary.
Time Frame: At the end of the Steep trendelenburg position, an average of 1 hour
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Number analyzed (Participants) | 32 | 34
units on a scale | 4.0 [3.0 to 5.0] | 3.0 [2.0 to 5.0]

3. Other Pre Specified Outcome: Post-operative Nausea
Time Frame: During 24hours after operation
Measure: Number; unit: events
Arm/Group | Moderate Neuromuscular Blockade (Moderate NMB Group) | Deep Neuromuscular Blockade (Deep NMB Group)
Number analyzed (Participants) | 32 | 34
events | 4 | 1

4. Other Pre Specified Outcome: Incidence of Residual Neuromuscular Blockade
Time Frame: During 24hours after operation
Measure: Number; unit: participants
Arm/Group | Moderate Neuromuscular Blockade (Moderate NMB Group) | Deep Neuromuscular Blockade (Deep NMB Group)
Number analyzed (Participants) | 32 | 34
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Moderate Neuromuscular Blockade | Deep Neuromuscular Blockade
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No